CLINICAL TRIAL: NCT02222389
Title: P20 Research Project 1 Contingency Management for the Treatment of Co-Occurring Alcohol and Drug Misuse
Brief Title: Contingency Management for the Treatment of Co-Occurring Alcohol and Drug Misuse
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Washington State University (Other)
Responsible Party: Principal Investigator, Michael McDonell, Associate Director & Associate Professor, Washington State University
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Treatment
Other Study IDs: 13210-001
Record Dates: First submitted 2014-07-22; First posted 2014-08-21 (Estimated); Last update posted 2018-09-18 (Actual); Status verified 2018-09

CONDITIONS: Co-Occurring Alcohol and Drug Misuse
MeSH Terms: conditions — Drug Misuse | interventions — Ethanol; Pharmaceutical Preparations

ARMS (4):
- CM for alcohol (Experimental): CM for alcohol
  Interventions: Behavioral: CM for Alcohol
- CM for drugs (Experimental): CM for drugs
  Interventions: Behavioral: CM for drugs
- CM for both substances (Experimental): CM for both substances
  Interventions: Behavioral: CM for both substances
- Non-Contingent group (Other): No CM for either substance, the Non-Contingent (NC) group
  Interventions: Behavioral: Non-Contingent group

INTERVENTIONS:
Behavioral: CM for Alcohol — Escalating reinforcement for alcohol abstinence.
  Alcohol-negative CM Participants draw chips out of a bowl containing 500 chips. Fifty percent of the chips will say "good job!" or a similar encouraging phrase, 41.8% of the chips will result in a small prize, 8% will result in a large prize, and 0.2% will result in a jumbo prize.
  Arms: CM for alcohol
Behavioral: CM for drugs — Escalating reinforcement for drug abstinence.
  Drug-negative participants will be invited to draw chips out of a bowl containing 500 chips. Fifty percent of the chips will say "good job!" or a similar encouraging phrase, 41.8% of the chips will result in a small prize, 8% will result in a large prize, and 0.2% will result in a jumbo prize.
  Arms: CM for drugs
Behavioral: CM for both substances — Escalating reinforcement for drug and alcohol abstinence.
  Drug- and alcohol-negative participants will be invited to draw chips out of a bowl containing 500 chips. Fifty percent of the chips will say "good job!" or a similar encouraging phrase, 41.8% of the chips will result in a small prize, 8% will result in a large prize, and 0.2% will result in a jumbo prize.
  Arms: CM for both substances
Behavioral: Non-Contingent group — Compensation for Non-Contingent control group participants is dependent only on providing urine samples, regardless of whether the urine tests are negative for alcohol and/or drugs.
  Arms: Non-Contingent group

SUMMARY:
Contingency management (CM) is a type of treatment used in the substance abuse field. Patients' behaviors are rewarded for adherence to a treatment plan. As an approach to treatment, contingency management emerged from the behavior therapy traditions in mental health. By most evaluations, contingency management procedures produce one of the largest effect sizes out of all mental health and educational interventions.

The purpose of this study is to perform a randomized, controlled trial to evaluate the ability of a culturally-tailored contingency management (CM) intervention to increase alcohol and drug abstinence among American Indian (AI) tribal members from two rural reservations in the Northwest.

ELIGIBILITY:
Inclusion Criteria:

1. Self-identify race as American Indian (AI)
2. Are seeking alcohol dependence and drug abuse treatment at a participating reservation
3. Are age 18 or older
4. Meet criteria of DSM-IV diagnosis of current alcohol dependence
5. Current drug misuse
6. Are not pregnant or planning to become pregnant for the duration of the study
7. Are English speaking
8. Have the ability to provide written informed consent

Exclusion Criteria:

1. Have significant risk of dangerous alcohol withdrawal, defined as a history of alcohol detoxification or seizure during the last 12 months AND expression of concern by the patient and/or healthcare provider
2. Meet criteria for DSM-IV diagnosis of drug dependence
3. Have significant risk of dangerous drug withdrawal and/or self-reported or medically documented severe withdrawal from drugs in the last 6 months
4. Have any medical or psychiatric condition, such as organic brain disorder, dementia, or psychotic disorder, that the Principal Investigator determines would compromise safe study participation
5. Are receiving drugs under the direction of a physician for pain management or another medical condition for which drug abstinence is contraindicated

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2015-06-01 (Actual); Primary Completion 2018-09-10 (Actual); Study Completion 2018-09-10 (Actual)

PRIMARY OUTCOMES:
Biochemically verified alcohol and/or drug abstinence | 24 weeks
  At every study visit, urine samples will be collected and analyzed for ethyl glucuronide and drugs. This helps assess Contingency Management as a treatment for alcohol and/or drug dependence.

SECONDARY OUTCOMES:
Self- reported data on alcohol and drug use | 24 weeks
  Measures used for self-reported data on alcohol and drug use:
  1. The Alcohol and Drug Timeline Follow Back (TLFB)
  2. The Current Opioid Misuse Measure (COMM)
  3. The Addiction Severity Index, Native American Version (ASI-NAV)
Other substance use | 24 weeks
  Amphetamine, methamphetamine, cocaine, and marijuana, will be measured by the same procedures described for urine tests of alcohol and drug metabolites.
Self- reported data on health behaviors | 24 weeks
  We will also collect secondary outcome data on health behaviors that frequently correlate with alcohol and drug misuse with the following measures:
  1. The Timeline Follow Back will be used to assess daily number of cigarettes smoked.
  2. Brief HIV Risk Behavior Scale
  3. Veteran's Rand- 12
  4. Self-Report Services Utilization Assessment

OTHER OUTCOMES:
Measures used for descriptive purposes and to assess success of randomization. | 24 weeks
  We will measure psychopathology with the Brief Symptom Inventory, a self-report instrument that will assess levels of anxiety, depression, impulsiveness, at baseline to characterize the psychiatric severity of the sample that has been used in previous studies of American Indians.
Measures used for descriptive purposes and to assess success of randomization. | 24 weeks
  The Fagerström Test of Nicotine Dependence will measure the presence and severity of nicotine dependence.
Measures used for descriptive purposes and to assess success of randomization | 24 weeks
  Interest in alcohol and drug abstinence will be assessed by the Stages of Change Readiness and Treatment Eagerness Scale.
Measures used for descriptive purposes and to assess success of randomization | 24 weeks
  In addition, other demographic, cultural, and cigarette smoking and alcohol use measures will be administered at baseline. These measures are part of the P20 Center Core measures. These measures include the Veteran's Rand-12 (already gathered as part of this study's protocol), the Behavioral Risk Factor Surveillance System Alcohol Survey, and demographic, cultural, and smoking behaviors (Behavioral Health Cooperative, Core Measures).

CONTACTS AND LOCATIONS:
Overall Officials: Mike McDonell, PhD, Principal Investigator — Washington State University
Locations (1):
- Washington State University, Spokane, Washington, United States

REFERENCES:
- [Derived] McDonell MG, Skalisky J, Burduli E, Foote A Sr, Granbois A, Smoker K, Hirchak K, Herron J, Ries RK, Echo-Hawk A, Barbosa-Leiker C, Buchwald D, Roll J, McPherson SM. The rewarding recovery study: a randomized controlled trial of incentives for alcohol and drug abstinence with a rural American Indian community. Addiction. 2021 Jun;116(6):1569-1579. doi: 10.1111/add.15349. Epub 2021 Jan 14. PMID 33220122